CLINICAL TRIAL: NCT07277777
Title: A Prospective, Randomized, Open-Label, Parallel-Group Clinical Trial Evaluating the Efficacy and Safety of 125I Seed Interstitial Brachytherapy Combined With Immune Checkpoint Inhibitor Therapy in Patients With Primary, Recurrent, or Metastatic Malignant Tumors Compared With Immune Checkpoint Inhibitor Therapy Alone
Brief Title: 125I Seed Brachytherapy Combined With Immunotherapy for Primary, Recurrent, or Metastatic Malignant Tumors
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Li Min (Other)
Responsible Party: Sponsor-Investigator, Li Min, Vice Director, Jinan Military General Hospital
Organization: Jinan Military General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 960HP20251119
Record Dates: First submitted 2025-11-30; First posted 2025-12-11 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Malignant Tumors
Keywords: lodine-125 Seed Brachytherapy; Immune Checkpoint Inhibitors; Local-Systemic Synergy; Recurrent or Refractory Tumors
MeSH Terms: conditions — Neoplasms; Recurrence | interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Intervention Model Description: This is a two-arm, parallel-group, phase II trial in which eligible patients with recurrent or refractory, unresectable malignant tumors are randomized in a 1:1 ratio to receive either 125I seed interstitial brachytherapy combined with immune checkpoint inhibitor therapy or immune checkpoint inhibitor therapy alone. Treatment allocation remains fixed throughout the study; no crossover between arms is planned. Patients will be treated and followed according to the assigned arm until disease progression, unacceptable toxicity, withdrawal of consent, or study completion.
Masking Description: Due to the procedural nature of 125I seed implantation, blinding of participants and treating clinicians is not feasible. However, imaging evaluators-including independent radiologists and nuclear medicine physicians responsible for tumor response assessment and imaging-based efficacy evaluations-will remain blinded to treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 125I Seed Brachytherapy + Immunotherapy (Experimental): Participants in this arm will receive CT-guided 125I seed interstitial brachytherapy, followed by systemic immune checkpoint inhibitor (ICI) therapy administered according to the approved dosing schedule for the selected agent. Seed implantation will be planned and delivered using standardized TPS-based dosimetric protocols, and immunotherapy will continue until progression, unacceptable toxicity, or study completion.
  Interventions: Drug: Immune Checkpoint Inhibitors; Other: 125I Seed Implantation
- Immunotherapy Alone (Active Comparator): Participants in this arm will receive systemic immune checkpoint inhibitor (ICI) therapy alone, following the same agent, schedule, and supportive care standards used in the experimental arm. No local radiotherapy or seed implantation will be performed. Treatment will continue until disease progression, unacceptable toxicity, or study completion.
  Interventions: Drug: Immune Checkpoint Inhibitors

INTERVENTIONS:
Drug: Immune Checkpoint Inhibitors — Examples include PD-1/PD-L1 inhibitors (e.g., pembrolizumab, nivolumab, camrelizumab, sintilimab) Administered per standard dosing schedule (e.g., every 2-3 weeks)
  Arms: 125I Seed Brachytherapy + Immunotherapy
Other: 125I Seed Implantation — PET/CT-guided implantation or CT-guided implantation Dose planning: D90 typically 90-140 Gy (adjusted per tumor type and size) Post-implant dosimetry: D90, V100, V150 recorded
  Arms: 125I Seed Brachytherapy + Immunotherapy
Drug: Immune Checkpoint Inhibitors — Same agent class and dosing schedule as the experimental arm Administered until disease progression, unacceptable toxicity, or study completion
  Arms: Immunotherapy Alone

SUMMARY:
This prospective randomized trial evaluates the efficacy and safety of combining 125I seed interstitial brachytherapy with immune checkpoint inhibitor therapy in patients with primary, recurrent, or metastatic malignant tumors. Immunotherapy has become an important systemic treatment option, yet many patients experience limited benefit due to low tumor immunogenicity, insufficient T-cell infiltration, and an immunosuppressive tumor microenvironment.

125I seed brachytherapy provides continuous low-dose-rate radiation to the tumor, promoting antigen release, enhancing dendritic cell activation, and potentially converting immunologically "cold" tumors into more responsive "hot" lesions. Integrating localized radiation with systemic immunotherapy may improve tumor response, prolong progression-free survival, and reduce recurrence.

Patients will be randomized 1:1 to receive 125I seed implantation plus immunotherapy or immunotherapy alone. The primary endpoints are objective response rate (ORR) and progression-free survival (PFS). Secondary endpoints include failure-free survival (FFS), overall survival (OS), disease control rate (DCR), duration of response (DoR), local control, recurrence rate, adverse events, and quality of life. Exploratory analyses will assess radiomics features, subgroup responses, and different patterns of recurrence. This study aims to determine whether adding 125I seed brachytherapy enhances the clinical benefits of immunotherapy across diverse malignant tumors.

DETAILED DESCRIPTION:
Patients with malignant tumors-including primary, recurrent, and metastatic disease-often exhibit heterogeneous responses to immune checkpoint inhibitors (ICIs). Limited tumor antigen exposure, poor immune infiltration, and an immunosuppressive tumor microenvironment frequently restrict the efficacy of immunotherapy. Strategies capable of enhancing local tumor immunogenicity and promoting systemic immune activation may improve clinical outcomes.

125I seed interstitial brachytherapy delivers continuous low-dose-rate radiation precisely to the tumor, offering both durable local control and immunomodulatory effects. Low-dose-rate irradiation can induce immunogenic tumor cell death, increase tumor antigen presentation, enhance dendritic cell activation, and promote T-cell recruitment. This process may convert immunologically inactive ("cold") tumors into immunologically active ("hot") lesions, thereby synergizing with ICIs to enhance anti-tumor immunity. Combining these modalities may improve objective response, delay treatment failure, reduce recurrence, and prolong survival.

This prospective, randomized, open-label, parallel-group trial will compare 125I seed brachytherapy plus immunotherapy with immunotherapy alone. Eligible patients will be randomized 1:1. The combination arm will receive CT-guided seed implantation followed by ICI therapy; the control arm will receive ICI monotherapy. All patients will undergo standardized imaging and clinical evaluations at pre-defined intervals.

The primary endpoints are objective response rate (ORR) and progression-free survival (PFS). Secondary endpoints include failure-free survival (FFS), overall survival, disease control rate, duration of response, local control rate, tumor recurrence rate, treatment-related and immune-related adverse events, and patient-reported quality of life. Exploratory analyses will investigate radiomics features associated with response, patterns of recurrence (local, regional, or distant), and subgroup differences across tumor types, disease stages, biomarker profiles, and treatment characteristics. These analyses may help identify imaging or clinical predictors of benefit, refine patient selection, and support biomarker-driven optimization of 125I seed brachytherapy combined with immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 80 years.
* Histologically or clinically confirmed primary, recurrent, or metastatic malignant tumor.
* At least one measurable lesion according to RECIST 1.1 or iRECIST.
* Tumor site suitable for 125I seed implantation under CT or PET/CT guidance.
* Planned to receive or eligible to receive an immune checkpoint inhibitor (ICI).
* ECOG performance status 0-2.
* Adequate organ function:

ANC ≥ 1.5 × 10⁹/L Platelets ≥ 80 × 10⁹/L Hemoglobin ≥ 90 g/L AST/ALT ≤ 3 × ULN (≤ 5 × ULN for liver metastasis) Creatinine clearance ≥ 50 mL/min

* Life expectancy ≥ 3 months.
* Ability to understand and sign informed consent.

Exclusion Criteria:

* Prior I-125 seed implantation at the planned treatment site.
* Active uncontrolled infection or systemic inflammatory disease.
* Known history of autoimmune disease requiring systemic immunosuppression.
* Prior treatment with immune checkpoint inhibitors within the last 4 weeks.
* Uncontrolled coagulopathy or contraindication to interventional seed implantation:

INR > 1.5 Platelets < 50 × 10⁹/L

* Tumor location that poses unacceptable procedural risk, including inability to obtain a safe puncture path.
* Severe cardiopulmonary dysfunction (e.g., heart failure, unstable arrhythmia, severe COPD).
* Pregnancy or breastfeeding.
* Known allergy or contraindication to radiopharmaceuticals, contrast agents, or anesthesia agents used during implantation.
* Any condition that, in the investigator's judgment, makes the participant unsuitable for the study (e.g., poor compliance, severe psychiatric disorder).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Every 6-12 weeks, up to 24 months
  Proportion of patients achieving complete response (CR) or partial response (PR) as defined by RECIST 1.1 or iRECIST, assessed via CT/MRI/PET-CT.
Progression-Free Survival (PFS) | Up to 24 months
  Time from randomization to radiographic disease progression or death from any cause.

SECONDARY OUTCOMES:
Failure-Free Survival (FFS) | Up to 24 months
  Time from randomization to the first occurrence of treatment failure, including disease progression, local recurrence, distant metastasis, discontinuation due to adverse events, or death.
Overall Survival (OS) | Up to 36 months
  Time from randomization to death from any cause.
Disease Control Rate (DCR) | Every 6-12 weeks, up to 24 months
  Percentage of patients achieving CR, PR, or stable disease (SD), according to RECIST 1.1/iRECIST.
Duration of Response (DoR) | Up to 24 months
  Time from first documentation of CR/PR until radiographic progression or death.
Local Control Rate (LCR) | Up to 24 months
  Proportion of treated lesions without local progression, based on imaging (CT/MRI/PET-CT) and dosimetric correlation of the implanted region.
Tumor Recurrence Rate | Up to 24 months
  Rate of local or regional tumor recurrence, defined by new lesions or regrowth within the same anatomical region as confirmed by imaging.
Treatment-Related Adverse Events (TRAEs) | From baseline until 90 days after last treatment
  Incidence, severity, and type of adverse events associated with treatment, graded according to CTCAE v5.0.
Immune-Related Adverse Events (irAEs) | Up to 24 months
  Incidence and grade of immunotherapy-related toxicities such as pneumonitis, colitis, dermatitis, endocrinopathies.
Quality of Life (QoL) | Baseline, Week 12, Week 24, and every 6 months up to 24 months
  Assessed using validated patient-reported instruments (e.g., EORTC QLQ-C30).

OTHER OUTCOMES:
Radiomics Features and Predictive Modeling | Up to 24 months
  Extraction of radiomic features from PET/CT or CT images to explore associations with ORR, PFS, recurrence pattern, and treatment response.
Subgroup Analyses | Up to 24 months
  Assessment of treatment effect by clinical subgroups (primary vs recurrent vs metastatic disease, tumor type, PD-L1 expression, inflammatory markers).
Patterns of Failure / Recurrence Patterns | Up to 24 months
  Classification of failure patterns (local, regional, distant) and correlation with dosimetry (D90, V100) and imaging biomarkers.

CONTACTS AND LOCATIONS:
Overall Officials: Min Li, Dr., Study Director
Locations (1):
- The 960th Hospital of People's Liberation Army (PLA), Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) will be made available to qualified researchers upon reasonable request after completion of the study and publication of the primary results. Data to be shared may include demographic information, treatment assignment, key efficacy outcomes, adverse events, and imaging-derived parameters. A data-sharing agreement will be required to ensure appropriate use of the dataset.
Supporting Information: Study Protocol, ICF
Time Frame: Individual participant data (IPD) will be available beginning 6 months after publication of the primary study results and will remain available for 5 years following publication, or until the main study database is closed, whichever occurs first.
Access Criteria: Qualified researchers affiliated with academic institutions or recognized research organizations may request access to de-identified individual participant data (IPD), including imaging-derived parameters, dosimetric results, and clinical outcome data.
  Requests must include a brief research proposal describing the scientific rationale, objectives, and planned analyses. Approval will be granted by the study's principal investigator and institutional ethics committee. Data will be shared through secure institutional data transfer systems after execution of a formal data sharing agreement that ensures patient confidentiality and compliance with applicable privacy regulations.